CLINICAL TRIAL: NCT01974544
Title: Prevention and Treatment Of Diabetes Complications With Gastric Surgery or Intensive Medicines
Acronym: PRODIGIES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-141
Record Dates: First submitted 2013-05-25; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
Keywords: diabetes complications; metabolic surgery; Intensive medicines
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Best medical treatment (Experimental): Fifty obese patients with kidney damage or high risk of kidney damage secondary to T2DM will will be treated using the American Diabetes Association protocol. Also this arm will be treated like: General interventions for all groups: blood presure, General interventions for all groups: dysilipidemia and General interventions for all groups: lifestyle establishes.
  Interventions: Drug: Best medical treatment; Drug: General interventions for all groups: blood presure; Drug: General interventions for all groups: dysilipidemia; Behavioral: General interventions for all groups: lifestyle
- gastric bypass surgery (Experimental): Fifty obese patients with kidney damage or high risk of kidney damage secondary to T2DM will undergo gastric bypass surgery, in the conventional procedure. Also this arm will be treated like: General interventions for all groups: blood presure, General interventions for all groups: dysilipidemia and General interventions for all groups: lifestyle establishes.
  Interventions: Procedure: gastric bypass; Drug: General interventions for all groups: blood presure; Drug: General interventions for all groups: dysilipidemia; Behavioral: General interventions for all groups: lifestyle
- sleeve gastrectomy (Experimental): Fifty obese patients with kidney damage or high risk of kidney damage secondary to T2DM will undergo sleeve gastrectomy surgery, in the conventional procedure. Also this arm will be treated like: General interventions for all groups: blood presure, General interventions for all groups: dysilipidemia and General interventions for all groups: lifestyle establishes.
  Interventions: Procedure: sleeve gastrectomy; Drug: General interventions for all groups: blood presure; Drug: General interventions for all groups: dysilipidemia; Behavioral: General interventions for all groups: lifestyle

INTERVENTIONS:
Drug: Best medical treatment — If patients are unable to maintain their haemoglobin A1c (HbA1c) values below 6.5% on diet alone, treatment with metformin 1g twice daily will be started. If HbA1c remains above 7.0% then liraglutide 0.6 mg once daily (with a subsequent increases to 1.2 mg and 1.8 mg once daily). If liraglutide is not tolerated then a Dipeptidyl peptidase IV inhibitor (sitagliptin, saxagliptin, linagliptin) or pioglitazone will be considered. If HbA1c remains above 7.5% long acting insulin analogues such as detemir o glargine will be added. If insulin is started liraglutide can be stopped. The insulin dose will be adjusted according to the morning fasting blood glucose concentration. Finally, Fast-acting meal time insulin (lispro, aspart or glulisine) will be added if glycemic goal is not achieved. Repaglinide can be considered in patients with significant renal impairment and in patients who refused insulin treatment.
  Other Names: Non surgical interventions; Glycemic control drugs
  Arms: Best medical treatment
Procedure: gastric bypass — For the gastric bypass, the gastric pouch will be adjusted to a volume of 15-20 ml. The alimentary limb will be a standard 150 cm and the biliopancreatic limb 50 cm. A hand-sewn gastro-jejunal anastomosis will be performed over a 34 French bougie
  Arms: gastric bypass surgery
Procedure: sleeve gastrectomy — The sleeve gastrectomy will be done using laparoscopic staplers over a 34 French bougie.The greater curvature will be dissected 4 cm proximal to the pylorus leaving the antrum. Short gastric vessels will be dissected using the harmonic scalpel up to the gastro-esophageal junction. The stapler will be reinforced. The resected stomach will be removed in a plastic bag through the left flank trocar
  Arms: sleeve gastrectomy
Drug: General interventions for all groups: blood presure — Patients will receive an angiotensin-converting-enzyme (ACE) inhibitor or angiotensin II receptor antagonists (ARA II) to meet strict blood pressure targets of the ADA / European Association for Study of Diabetes (EASD) or in the presence of micro or macroalbuminuria. In addition to ACE inhibitors (or if there were side-effects, an angiotensin-II receptor antagonist), calcium antagonist, diuretics or Beta blockers can be added as needed. Aspirin 100 mg daily will be used for secondary prevention in patients with a history of ischaemic cardiovascular disease.
  Other Names: Management elevated blood pressure in patients with T2DM
Drug: General interventions for all groups: dysilipidemia — Raised fasting serum cholesterol concentrations (greater than 4.5 mmol/L) or combined dyslipidaemias will be treated with atorvastatin 10-80mg once daily. Gemfibrozilo or fenofibrate once daily can be used for isolated hypertriglyceridaemia (fasting serum triglyceride concentration >4.0 mmol/L), or fenofibrate can be added to statin treatment if the fasting serum triglyceride concentration was also raised (>4.0 mmol/L).
  Other Names: Management of dyslipidemia
Behavioral: General interventions for all groups: lifestyle — Exercise is an important part of the diabetes management plan. The ADA recommendations for the adults with diabetes is at least 150 min/week of moderate-intensity aerobic physical activity (50-70% of maximum heart rate), with no more than two consecutive days without exercise. A kinesiologist will design an individual plan of physical training for each patient. Also, a nutritionist will be design an individual dietitian plan, this plan should be formulated as a collaborative therapeutic alliance among the patient and family, physician, and other members of the health care team.
  Other Names: Therapeutic lifestyle modification

SUMMARY:
The obesity and type 2 diabetes mellitus (T2DM) are among the most threatening health crisis for the 21st century. Currently, it is estimated that there are 205 million people with T2DM worldwide. Chile has a similar magnitude of problem with the prevalence of diabetes increasing from 6.3% in 2003 to 9.4% in 2010. T2DM is a complex disease characterized by hyperglycemia, insulin resistance and a relative β-cell failure. Well-known studies for the treatment of T2DM (ADVANCE trial) showed that intensive medical treatment significantly reduces the complication of diabetes. On the other hand, less than 40% of patients with T2DM achieve a metabolic control of diabetes, despite medical treatment. Recently, bariatric surgery has emerged as an effective treatment for T2DM. Data from different sources has shown that Roux-en-Y Gastric Bypass (RYGB) can place T2DM into remission. More recently, Sleeve Gastrectomy (SG) has been shown to also impact metabolically and hence also emerged as an attractive T2DM-controlling bariatric procedure with fewer complications than RYGB. Recently, the International Federation for Diabetes has supported the use gastrointestinal surgery initially developed for morbid obesity as an option to treat patients with diabetes. In the current proposal the investigators aim to address several issues concerning metabolic surgery and the ability of the most common bariatric procedures performed to control diabetes. The investigators are proposing a prospective randomized trial comparing RYGB, SG and the best medical treatment availed for the T2DM in poorly control patients with the primary endpoint being 36 month glycemic control (patients achieving HbA1C < 6.5%, normal glucose levels not requiring medication). The main working hypothesis is that RYGB and SG achieves better glycemic control than the best treatment availed for the T2DM based on more effective mechanisms to enhance insulin secretion, insulin sensitivity, lipid metabolism and blood pressure control. The goals are, 1) Is gastric bypass surgery and sleeve gastrectomy safe for the microvascular complications of T2DM?; 2) Can gastric bypass, sleeve gastrectomy surgery and intensive non surgical treatment reverse or reduce the progression of microvascular complications of T2DM?; and 3) Can gastric bypass and sleeve gastrectomy realize a return on investment within 2 years in patients with type 2 diabetes who are at risk of developing or deteriorating microvascular complications?

DETAILED DESCRIPTION:
Currently 205 million patients in the world suffer with Type 2 diabetes and severe and complex obesity. The obesity is defined as a body mass index above 30 kg/m2 with life or limb threatening co-morbidities.

The bariatric surgery increase in worldwide, but their effects on the microvascular complications of T2DM have never been the focus of a randomised controlled clinical trial.

To address this research question a three arms on randomised controlled clinical trial comparing gastric bypass surgery, sleeve gastrectomy and modern best medical care is required to investigate differences in long term glycaemia and microvascular complications of T2DM.

This is a prospective intervention study on patients with T2DM and obesity undergoing gastric bypass surgery, sleeve gastrectomy or non surgical best medical care. Patients will have T2DM for more than 2 years and have or be at high risk of developing kidney damage. Patients will be recruited from specialist medical and surgical clinics.

We expect to screen approximately 300 patients to allow 75 to be randomized. Twenty five subjects with kidney damage or high risk of kidney damage secondary to T2DM will undergo gastric bypass surgery. Another 25 sleeve gastrectomy and the final 25 will be treated using the American Diabetes Association protocol. Patients with HbA1c ≥9.0% will undergo individualised optimisation of glycaemia as this should improve surgical outcomes. Particular attention will be given to the avoidance of hypoglycaemia. Patients' other risk factors (including hypertension and dyslipidaemia) will be optimised based on the International Diabetes Federation guidelines.

The clinical endpoints that will be assessed are: renal function, peripheral and autonomic nervous system function, the retina, of direct healthcare cost, glycaemic control, blood pressure, lipids, quality of life, postprandial responses, treatment complications.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes with HbA1c > 7%
2. Duration of diabetes of more than 2 years
3. The glomerular filtration rate (GFR) > 30 ml/min per 1.73 m2
4. BMI < 35 kg/m2
5. Age 18-65
6. Established microalbuminuria or at high risk of microalbuminuria

Exclusion Criteria:

1. Type 1 diabetes or positive Glutamic acid decarboxylase antibodies (Anti-GAD)
2. BMI >35 kg/m2
3. End stage retinopathy, nephropathy or neuropathy (defined as high risk/advanced proliferative retinopathy on the Early Treatment Diabetic Retinopathy Study Severity Scale or blindness, Stage 5 chronic kidney disease, patients requiring dialysis or transplantation, Stage 3 peripheral neuropathy)
4. Unacceptably high risk for general anaesthesia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in the microvascular complications of type 2 diabetes, specifically diabetic kidney disease | baseline at 1 month before the intervention and 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36 month after intervention
  These outcome will be measured through the glomerular filtration rate (GFR), (MDRD-1 equation: GFR (expressed in ml/min/1.73 m2), and Albuminuria (ACR (mg/g).
Change in the microvascular complications of type 2 diabetes, specifically Retinopathy. | baseline at 1 month before the intervention, 12 y 24 month after intervention
  This will be measured through assessment by ophthalmologist.
Change in the microvascular complications of type 2 diabetes, specifically peripheral and sympathic neuropathy. | baseline at 1 month before the intervention, 12, 24 y 36 month
  This will be measured through assessment nerve conduction, sensory nerve conduction, motor nerve conduction, sympathic skin response.

SECONDARY OUTCOMES:
Assessment of the optimization of the metabolic control, defined by the International Diabetes Federation | baseline at 1 month before the intervention and 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36 month after the intervention
  This will be measured through haemoglobin A1c (HbA1c) (%), continuous glucose monitoring, blood pressure (mmhg), total cholesterol (mg/dL), HDL (mg/dL), LDL (mg/dL), triglycerides (mg/dL).
Assessment of treatment complications | 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36 month after intervention
  This will be measured through the record of all treatment complications like: Infection or surgical bleeding, inflammation of the veins for drug administration, temporary digestive disorders, gastroesophageal reflux disease, or acute retention of urine infection, prolonged pain in the area of operation. Specifically for the Gastric Bypass, intestinal fistulas poor healing of sutures, nutritional deficiencies, excessive weight loss. Less often marginal ulcerative lesions and intestinal obstruction. In the other side, the sleeve gastrectomy: dehiscence of the suture line and nutritional complications.
Assessment of the quality of life. | baseline at 1 month before the intervention and 3, 6, 12, and 24 month after the intervention
  This will be measured through the Diabetes Quality of Life Questionnaire.
Assessment of macrovascular events | baseline at 1 month before the intervention and 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36 month after the intervention
  This will be measured through the record of all macrovascular events, like cardiovascular deaths, nonfatal myocardial infarction, cardiovascular interventions, nonfatal stroke, amputation or surgery for peripheral atherosclerotic artery disease.
How many patients not requiring antidiabetic agents | baseline 1 month after intervention, and at 6, 12, 18, 24, 30, and 36 month after intervention
  This will be measured through the record of number of patient who requiring oral antidiabetic agent, number of patient who requiring insulin, and both.

CONTACTS AND LOCATIONS:
Overall Officials: Boza Camilo, MD surgeon, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile